CLINICAL TRIAL: NCT05624437
Title: BElimumab corticoSteroids Sparing Treatment in Systemic Lupus
Brief Title: BElimumab corticoSteroids Sparing Treatment in Systemic Lupus Erythematosus
Acronym: BESST
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier de Niort (Other)
Responsible Party: Principal Investigator, Perier, Doctor, Centre Hospitalier de Niort
Other Study IDs: CHNiort
Record Dates: First submitted 2021-11-29; First posted 2022-11-22 (Actual); Last update posted 2022-11-22 (Actual); Status verified 2022-11

CONDITIONS: SLE (Systemic Lupus)
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — Electronic Health Records

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: data record — data record

SUMMARY:
BELIMUMAB, anti-BLyS human monoclonal antibody, is the first immunotherapy used for the treatment of systemic lupus erythematosus (SLE) which was licensed in 2011 in France.

Currently, Belimumab is reimbursed for the treatment of active SLEwith autoantibody-positive after intolerant or initial failure of first-line traitment (anti malaria, non-steroidal anti-inflammatory drugs, glucocorticoids and/ou immunomodulatory agents).

EUropean League Against Rheumatism (EULAR) suggest the following terminology of "low dose" when steroids are less than 7.5 mg/day (prednisone equivalent) because this dose range is often used for maintenance therapy for many rheumatic diseases requiring glucocorticoids and it is relatively few adverse effects.

In patients with SLE, a significant proportion of the damage could be attributed to corticosteroid therapy, and this damage accumulated over time.

Thanks to randomised and subgroups trials, post-hoc analysis , BELIMUMAB seems to be interesting in the maintain of lowest possible dose of glucocorticoids. However, these studies were not design with this aim, so it is impossible to conclude.

Thus, BELIMUMAB seems to be very interesting treatment to redcuce glucocorticoids level.

We conduce a multicentric French study in real-life settings, to assess the ability of belimumab to achieve low-dose of steroids.

ELIGIBILITY:
Inclusion Criteria:

* person aged ≥ 18 years
* with SLE according to ACR/EULAR criteria 2019
* started treatment by BELIMUMAB between 13 / July / 2011 to 13 / July / 2020
* following in an hospital center in Poitiers, La Rochelle, Rochefort, Niort, Angoulême, Nantes, Rennes, Tours, Angers
* affiliate or beneficiary of a social security scheme

Exclusion Criteria:

* Persons Under guardianship or curatorship or without civil law
* Pregnant and breastfeeding
* Persons who refused to participate
* Patients who stoppped BELIMUMAB before 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: person aged ≥ 18 years
  * with SLE according to ACR/EULAR criteria 2019
  * started treatment by BELIMUMAB between 13 / July / 2011 to 13 / July / 2020
  * following in an hospital center in Poitiers, La Rochelle, Rochefort, Niort, Angoulême, Nantes, Rennes, Tours, Angers
  * affiliate or beneficiary of a social security scheme
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2021-11-19 (Actual); Primary Completion 2021-11-19 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
number of patients whith low dose of steroids at six months after BELIMUMAB | at six months after BELIMUMAB
  number of patients whith low dose of steroids at six months after BELIMUMAB

SECONDARY OUTCOMES:
number of patients whith low dose of steroids at 12, 18 and 24 months after BELIMUMAB | 12, 18 and 24 months after BELIMUMAB
  number of patients whith low dose of steroids at 12, 18 and 24 months after BELIMUMAB
cumulative dose of steroids at 6, 12, 18, 24 months | 6, 12, 18, 24 months
  cumulative dose of steroids at 6, 12, 18, 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- CH Niort, Niort, France

IPD SHARING:
Plan to Share IPD: Undecided